CLINICAL TRIAL: NCT04962204
Title: Efficacy of Virtual Visitation in Intensive Care Unit During COVID-19 Pandemic: Randomized Controlled Trial
Brief Title: Virtual Visitation in Intensive Care Unit Study
Acronym: ISEEU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Seung-Young Oh, Clinical Assistant Profeessor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2105-188-1224
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Critically Ill Patients
MeSH Terms: interventions — Physicians; Caregivers

STUDY DESIGN:
Intervention Model Description: Interventional group Control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual visitation group (Active Comparator): Virtual visits between patients-caregivers and virtual interviews between physicians-caregivers for 15minutes once a day
  Interventions: Behavioral: Virtual meeting between patients/physicians and caregiver
- Control group (No Intervention): Phone interview between physicians-caregivers once a day

INTERVENTIONS:
Behavioral: Virtual meeting between patients/physicians and caregiver — Virtual visits between patients-caregivers and virtual interviews between physicians-caregivers for 15minutes once a day
  Arms: Virtual visitation group

SUMMARY:
The purpose of this study is to identify the efficacy of virtual visitation in Intensive Care Unit on patients and their caregivers during COVID-19 Pandemic.

DETAILED DESCRIPTION:
After being informed about the study, all patients who meet the eligibility requirements will be randomized in a 1:1 ratio to intervention group (Virtual visitation once a day) or Control group (Phone interviews once a day).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are expected to stay in the intensive care unit for more than 48 hours
* Patients with a RASS score of -2 or higher

Exclusion Criteria:

* Patients who discharge or die within 48 hours of admission to ICU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
FS-ICU score from caregivers at discharge or 7 days after initiation of study enrolled | 7 days
  The FS-ICU survey score reflected the satisfaction degree of caregivers. The overall satisfaction score is derived from questions 1 through 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Woo HY, Oh SY, Lim L, Im H, Lee H, Ha EJ, Ryu HG. Efficacy of Virtual Visitation in ICU During COVID-19 Pandemic: The ICU Visits Randomized Controlled Trial. Crit Care Med. 2024 Dec 1;52(12):e593-e603. doi: 10.1097/CCM.0000000000006429. Epub 2024 Sep 16. PMID 39283178